CLINICAL TRIAL: NCT05395052
Title: A Phase I, Open-Label, Multicenter Study of FT536 as Monotherapy and in Combination With Monoclonal Antibodies in Subjects With Advanced Solid Tumors
Brief Title: FT536 Monotherapy and in Combination With Monoclonal Antibodies in Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was terminated by the Sponsor.
Sponsor: Fate Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FT536-101
Record Dates: First submitted 2022-05-13; First posted 2022-05-27 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Non Small Cell Lung Cancer; Colorectal Cancer; Breast Cancer; Ovarian Cancer; Pancreatic Cancer; Head and Neck Cancer; GastroEsophageal Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Breast Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms; Head and Neck Neoplasms | interventions — Cyclophosphamide; fludarabine; Influenza Vaccines; Interleukin-2; avelumab; pembrolizumab; Nivolumab; atezolizumab; Trastuzumab; Cetuximab; amivantamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort A/A2/AA/AA2: FT536 Monotherapy (Experimental): FT536 monotherapy in participants with locally advanced or metastatic non-small cell lung cancer (NSCLC), colorectal cancer (CRC), breast cancer (BC), ovarian cancer, or pancreatic cancer.
  Interventions: Drug: FT536; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: IL-2
- Cohort B/B2/BB/BB2: FT536 + Avelumab (Experimental): FT536 + avelumab combination therapy in participants with locally advanced or metastatic solid tumor indications with documented PD-L1 expression.
  Interventions: Drug: FT536; Drug: Cyclophosphamide; Drug: Fludarabine; Combination Product: Avelumab; Drug: IL-2
- Cohort C/C2/CC/CC2: FT536 + Pembrolizumab, Nivolumab, or Atezolizumab (Experimental): FT536 + pembrolizumab, nivolumab, or atezolizumab in participants with locally advanced or metastatic solid tumor indications with documented PD-L1 expression.
  Interventions: Drug: FT536; Drug: Cyclophosphamide; Drug: Fludarabine; Combination Product: Pembrolizumab; Combination Product: Nivolumab; Combination Product: Atezolizumab; Drug: IL-2
- Cohort D/D2/DD/DD2: FT536 + Trastuzumab (Experimental): FT536 + trastuzumab in participants with locally advanced or metastatic documented human epidermal growth factor receptor 2 (HER2+) expressing tumors
  Interventions: Drug: FT536; Drug: Cyclophosphamide; Drug: Fludarabine; Combination Product: Trastuzumab; Drug: IL-2
- Cohort E/E2/EE/EE2: FT536 + Cetuximab (Experimental): FT536 + cetuximab in participants with locally advanced or metastatic squamous NSCLC, CRC, or head and neck cancer.
  Interventions: Drug: FT536; Drug: Cyclophosphamide; Drug: Fludarabine; Combination Product: Cetuximab; Drug: IL-2
- Cohort F/F2/FF/FF2: FT536 + Amivantamab (Experimental): FT536 + amivantamab in participants with locally advanced or metastatic NSCLC.
  Interventions: Drug: FT536; Drug: Cyclophosphamide; Drug: Fludarabine; Combination Product: Amivantamab; Drug: IL-2

INTERVENTIONS:
Drug: FT536 — FT536 is an allogeneic natural killer (NK)-cell immunotherapy
  Other Names: NK Cell Therapy
Drug: Cyclophosphamide — Lympho-conditioning agent
  Other Names: Cy
Drug: Fludarabine — Lympho-conditioning agent
  Other Names: Flu
Drug: IL-2 — For Cohort AA ONLY: To be combined with FT536 at the MTD or MAD
  Other Names: Interleukin-2
  Arms: Cohort A/A2/AA/AA2: FT536 Monotherapy
Combination Product: Avelumab — Monoclonal antibody
  Other Names: Bavencio
  Arms: Cohort B/B2/BB/BB2: FT536 + Avelumab
Combination Product: Pembrolizumab — For Cohorts C/CC, the combination product (monoclonal antibody) will be ONE of the following: pembrolizumab, nivolumab, or atezolizumab.
  Other Names: Keytruda
  Arms: Cohort C/C2/CC/CC2: FT536 + Pembrolizumab, Nivolumab, or Atezolizumab
Combination Product: Nivolumab — For Cohorts C/CC, the combination product (monoclonal antibody) will be ONE of the following: pembrolizumab, nivolumab, or atezolizumab.
  Other Names: Opdivo
  Arms: Cohort C/C2/CC/CC2: FT536 + Pembrolizumab, Nivolumab, or Atezolizumab
Combination Product: Atezolizumab — For Cohorts C/CC, the combination product (monoclonal antibody) will be ONE of the following: pembrolizumab, nivolumab, or atezolizumab.
  Other Names: Tecentriq
  Arms: Cohort C/C2/CC/CC2: FT536 + Pembrolizumab, Nivolumab, or Atezolizumab
Combination Product: Trastuzumab — Monoclonal antibody
  Other Names: Herceptin
  Arms: Cohort D/D2/DD/DD2: FT536 + Trastuzumab
Combination Product: Cetuximab — Monoclonal antibody
  Other Names: Erbitux
  Arms: Cohort E/E2/EE/EE2: FT536 + Cetuximab
Combination Product: Amivantamab — Monoclonal antibody
  Other Names: Rybrevant
  Arms: Cohort F/F2/FF/FF2: FT536 + Amivantamab
Drug: IL-2 — For Cohorts BB-FF ONLY: To be combined with FT536 + mAb at the MTD or MAD
  Other Names: Interleukin-2
  Arms: Cohort B/B2/BB/BB2: FT536 + Avelumab; Cohort C/C2/CC/CC2: FT536 + Pembrolizumab, Nivolumab, or Atezolizumab; Cohort D/D2/DD/DD2: FT536 + Trastuzumab; Cohort E/E2/EE/EE2: FT536 + Cetuximab; Cohort F/F2/FF/FF2: FT536 + Amivantamab

SUMMARY:
This is a Phase 1 dose-finding study of FT536 given in combination with a monoclonal antibody following lymphodepletion in participants with advanced solid tumors. The study will consist of a dose-escalation stage and an expansion stage where participants will be enrolled into indication-specific cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Participants with locally advanced or metastatic disease who have progressed/relapsed, are refractory, intolerant to or refuse standard therapy approved for their specific tumor type:

Cohort A/A2/AA/AA2: NSCLC, CRC, BC, ovarian cancer, or pancreatic cancer

Cohorts B/B2/BB/BB2 and C/C2/CC/CC2: Subjects with NSCLC, HNSCC, gastroesophageal adenocarinoma, triple negative breast cancer, or urothelial carcinoma whose tumors express PD-L1 according to defined cutoff

Cohort D/D2/DD/DD2: Subjects with advanced solid tumor whose tumor(s) express HER2 defined as: ≥2+ by IHC, Average HER2 copy number ≥4 signals per cell by in situ hybridization or ≥4 copies as determined by next generation sequencing

Cohort E/E2/EE/EE2: Squamous NSCLC; head and neck cancer that relapsed or progressed following prior cetuximab treatment; CRC subjects who are KRAS/NRAS/BRAF wild-type are required to have progressed/relapsed on prior cetuximab or panitumumab

Cohort F/F2/FF/FF2: NSCLC known to have at least one of the following: epidermal growth factor receptor (EGFR) driver mutation(s) and have progressed on or were intolerant to at least one prior line of EGFR Tyrosine Kinase Inhibitor (TKI) or were not candidates for or declined TKI; mesenchymal-epithelial transition (MET) exon 14 skipping mutation that has progressed on or intolerant of at least one prior line of MET TKI or were not candidates for or declined TKI; MET amplification defined as MET/CEP7 ratio ≥1.8 by Fluorescence in situ hybridization (FISH)

* Has measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* For subjects with >1 measurable lesion by RECIST v1.1 that can be safely accessed, willingness to undergo tumor biopsy
* Agrees to contraceptive use for women and men as defined in the protocol

Exclusion Criteria:

* Is a pregnant or breast-feeding female
* Has Eastern Cooperative Oncology Group (ECOG) performance status ≥2
* Has evidence of insufficient organ function
* Has clinically significant cardiovascular disease including left-ventricular ejection fraction < 45%
* Has received any therapy within 2 weeks prior to Day 1 or five half-lives, whichever is shorter or any investigational therapy within 28 days prior to Day 1
* Has a known active malignancy in the central nervous system (CNS) that hasn't remained stable for at least 3 months following effective treatment for CNS disease
* Has a non-malignant CNS disease such as stroke, epilepsy, CNS vasculitis or neurodegenerative disease or receipt of medications for these conditions
* Has had any active malignancy other than those studied in this trial within 2 years of the first dose of study therapy
* Is currently receiving or likely to require immunosuppressive therapy
* Has an active bacterial, fungal, or viral infections including hepatitis B, hepatitis C, or human immunodeficiency virus (HIV)
* Has received a live vaccine within 6 weeks prior to start of lympho-conditioning
* Has a known allergy to albumin (human) or dimethyl sulfoxide (DMSO)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2023-08-11 (Actual); Study Completion 2023-08-11 (Actual)

PRIMARY OUTCOMES:
Determine the Recommended Phase 2 Dose (RP2D) | Up to approximately 3 years
  The RP2Ds of FT536 monotherapy and FT536 + monoclonal antibody (mAbs) will be determined. The RP2D will be determined based on the overall safety and efficacy profile.
Number of Participants with ≥ Adverse Event (AE) according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), v5.0 | Following enrollment completion within dose escalation and expansion, approximately 3 years
  The safety and tolerability of FT536 monotherapy and in combination with mAbs will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Fate Trial Disclosure, Study Director — Fate Therapeutics
Locations (5):
- United States (5):
  - Honor Health Research Institute, Scottsdale, Arizona
  - UCLA Division of Hematology-Oncology, Los Angeles, California
  - Hackensack University Medical Center - John Theurer Cancer Center, Hackensack, New Jersey
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - NEXT Oncology, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No